CLINICAL TRIAL: NCT06917703
Title: Effectiveness of a Mobile Health Program on Blood Glucose and Gestational Weight Gain in Pregnant Women: A Mixed-Methods Study
Brief Title: Effectiveness of a Mobile Health Program in Pregnant Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Tzu-Ling Chen, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: (1154)114A-12; CHGH113-IU02 (Registry Identifier: Effectiveness)
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy; Gestational Age and Weight Conditions; Eating Behaviors; Literacy; E-learning
Keywords: pregnancy; health literacy; E-learning; gestational weight gains; nutriention
MeSH Terms: conditions — Feeding Behavior; Literacy

STUDY DESIGN:
Intervention Model Description: To assess the effectiveness of the i-PregMom mobile application and digital dietary image recording on blood glucose control and gestational weight gain, a randomized controlled design with a double repeated measures approach will be conducted (Intervention group: n=80; Control group: n=80). Data will be collected at three time points:
  * Baseline (10-14 weeks of gestation)
  * Two weeks post-intervention (12-16 weeks of gestation)
  * Three months post-intervention (24-28 weeks of gestation) The intervention group will receive face-to-face nutrition education (15-30 min/session) based on the Health Promotion Administration's pregnancy dietary guidelines and access to the i-PregMom mobile application for continuous dietary management. The control group will receive only face-to-face nutrition education (15-30 min/session) based on standard pregnancy dietary guidelines.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Health Program (Experimental): The intervention group will receive face-to-face nutrition education (15-30 min/session) based on the Health Promotion Administration's pregnancy dietary guidelines and access to the i-PregMom mobile application for continuous dietary management.
  Interventions: Other: E-learning
- rountine care (No Intervention): The control group will receive only face-to-face nutrition education (15-30 min/session) based on standard pregnancy dietary guidelines.

INTERVENTIONS:
Other: E-learning — in experience group
  Arms: Mobile Health Program

SUMMARY:
1. To evaluate the usability and user experience of the i-PregMom mobile application and digital dietary image recording among pregnant women.
2. To examine the effectiveness of digital mobile health interventions on blood glucose levels and gestational weight gain among pregnant women from 10-14 weeks to 24-28 weeks of gestation.

DETAILED DESCRIPTION:
1. Sociodemographic variables: age, education level, marital status, occupation, and socioeconomic status.
2. Obstetric variables: gravidity, history of miscarriage, pregnancy complications, and mode of delivery.
3. Pre-pregnancy BMI.
4. Dietary habits, perceived healthy eating behaviors, and dietary patterns.
5. Psychological distress and depressive symptoms.
6. Gestational blood glucose levels and GWG

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women aged ≥18 years.

Singleton pregnancy.

Pregnant women between 10 and 14 weeks of gestation, with gestational age calculated based on the first day of the last menstrual period.

Able to listen, speak, read, and write in Chinese.

Willing to provide prenatal weight and blood glucose data.

Possess a mobile communication device (such as a smartphone or social media account) and be able to receive emails.

Exclusion Criteria:

* Engaged in weight loss activities prior to pregnancy.

Diagnosed with chronic illnesses that may affect weight changes (e.g., psychiatric disorders, thyroid diseases).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Gestational Weight Gain in Pregnant | o Gestational Weight Gain (GWG) will be recorded three times (10-14, 12-16, and 24-28 weeks of gestation) based on maternity health records to analyze trends in weight changes and the impact of the mobile health intervention.
  Gestational Weight Gain (GWG) will be recorded three times (10-14, 12-16, and 24-28 weeks of gestation) based on maternity health records to analyze trends in weight changes and the impact of the mobile health intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- 365, Ming-Te Rd, Peitou District, Taipei 11219, Taiwan, ROC, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data will be anonymized and used solely for analysis in preparation for publication; it will not be shared."